CLINICAL TRIAL: NCT03730636
Title: Procalcitonin and Duration of AntiBiotherapy In Late Onset Sepsis of Neonate
Acronym: PROABIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P170928J; 2018-AO1396-49 (Other: ANSM)
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-03

CONDITIONS: Sepsis
Keywords: Late Onset Sepsis (LOS); antibiotic therapy duration; procalcitonin (PCTR)
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCT-guided strategy (Experimental): Measurement of PCT concentration will be performed every two days and the ATB therapy will be stopped when PCT level reaches a value equal or below 0.5ng/mL.
  Interventions: Procedure: PCT dosage
- Usual practice (control group) (No Intervention): Management of LOS and treatment is based on the attending clinician's practice and according to the usual practice.

INTERVENTIONS:
Procedure: PCT dosage — Measurement of PCT concentration will be performed every two days and the ATB therapy will be stopped when PCT level reaches a value equal or below 0.5ng/mL.
  Arms: PCT-guided strategy

SUMMARY:
The duration of antibiotic (ATB) therapy in late onset sepsis (LOS) of the neonate is currently not based on scientific data. The current PROABIS trial will study the use of a biological marker, procalcitonin (PCT), to guide ATB therapy duration in neonates with LOS.

Our hypothesis is that the use of procalcitonin guidance can reduce of 30% the duration of ATB treatment without increasing recurrence of infection and mortality.

DETAILED DESCRIPTION:
Randomized controlled multicenter open trial comparing the efficacy of PCT guided strategy (superiority aspect) and safety (non-inferiority aspect) versus usual strategy in LOS of the neonate.

After inclusion, patients are randomly assigned (in a 1:1 ratio) to duration of ATB therapy according to PCT guidance (experimental group) or to standard of care (control group).

Experimental group:

For patients randomly assigned in the PCT-guided group, a PCT concentration is measured at D0 (randomisation), at D2 and then, every two days until PCT value is equal or below 0.5 ng/mL.

The physician in charge of the neonate will be strongly encouraged to stop ATB treatment as soon as the PCT value is equal or below 0.5 ng/mL.

Control group:

In the control group, management of LOS and treatment are based on the attending clinician's practice and according to the usual practice (No PCT dosage).

In both groups data will be collected at the follow-up visit (day 14±2 after randomization) or the day of discharge from the hospital (if before 14±2 days) and at the end of the study visit (day 28± 2 after randomization) In case of transfer to another service or hospital or known re hospitalization before day28, outcomes will be collected from the service receiving the patient.

A phone call will be made to the parents, only in case of discharge before 28 days. following randomization. This phone call will be made 28± 2 days after randomization to identify adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born at 24 or more weeks of gestation,
* Aged over 96 hours of life, i.e. from the 5th day of life and less than 45 gestational weeks at diagnosis of assumed or proven LOS,
* Weight at the inclusion ≥ 700 g,
* Treated by ATB therapy for less than 48 hours,
* When the physician decides to continue de empiric ATB treatment beyond the initial 48-h period,
* Written informed consent signed by both parents (in the absence of one of the two parents the day of inclusion, the new born can be included with the signature of only one parent.The second parent must give oral consent and sign the consent form as soon as possible "before day 28"),
* Affiliation to a social security system (recipient or assign).

Exclusion Criteria:

* Neonates with non-indication of ATB treatment following the 48h-initial empiric period.
* ATB treatment within the 48h before the current episode of infection; except for taking antibiotics for prophylactic purposes (ex: digestive decontamination), pulmonary-targeted treatments for atypical germs and antibiotics by local means (ex.: eye drops).
* Patients diagnosed with severe infections (meningitis and/or septic shock) or needing prolonged therapy (ex: endocarditis, bone infection, deep seated infection, abscesses). Septic shock is defined by fluid resistant hypotension requiring vasopressor therapy.
* Infections not contracted during the hospitalization in the neonatal period or revealed more than 48 hours after hospital discharge.
* Neonates during treatment by extracorporeal membrane oxygenation or extra-corporeal circulation, and within the 72h after the end of the treatment.
* Neonates previously included in the Proabis study.
* Participation with another interventional study involving human subjects or being in the exclusion period at the end of a previous study involving human subjects.

Ages: 96 Hours to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 511 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of the PCT guided ATB strategy on the duration of ATB treatment compared to usual ATB strategy | up to 28 days
  Number of days between start and end of treatment, including treatment of the recurrence, if any

SECONDARY OUTCOMES:
Non-inferiority of the PCT-guided ATB strategy to usual strategy on mortality at 28 days following randomization | 28 days
  Mortality rate at 28 days following randomization
Non-inferiority of the PCT-guided ATB strategy to usual strategy on recurrence of infection within 72 hours after ending ATB therapy. | 28 days
  Proportion of infants with a treatment failure and recurrence of infection within 72h after ending ATB treatment and requiring additional course of ATBs.
Description on the total number of assumed or proven bacterial infections within the 28 days following randomization. | 28 days
  Total number of assumed or proven bacterial infections within the 28 days following randomization, excluding the primary infection and its recurrence
To compare the cumulative dose of received ATB treatment (mg/kg). | Day 28
  Cumulative dose of ATB treatment (mg/kg), defined as the total dose (in mg/kg) between start and end of treatment, including treatment of the recurrence, if any
To describe the bacteriological epidemiology of LOS | 28 days
  Recording of all the bacteriological species identified in blood or other samples during the LOS
Proportion of patients with bronchopulmonary dysplasia | 28 days
  Proportion of patients with bronchopulmonary dysplasia in order to assess the proportion of patients with bronchopulmonary dysplasia at 28 days
Proportion of patients with at least one event between randomization and day 28 among death, recurrence of infection and bronchopulmonary dysplasia. | 28 days
  Proportion of patients with at least one event between randomization and day 28 among death, recurrence of infection and bronchopulmonary dysplasia in order to evaluate the endpoint combining death or recurrence of infection or bronchopulmonary dysplasia
Antibiotics free days at D28 | 28 days
  Antibiotics free days at D28is defined as the number of days alive without any antibiotics at day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine MITANCHEZ, PU-PH, Principal Investigator — Department of Neonatology Bretonneau Hospital
Locations (1):
- Department of Neonatology Bretonneau Hospital, Paris, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided